CLINICAL TRIAL: NCT05216107
Title: Predicting Morbidity and Mortality in Elderly Surgical Patients: Prospective Multicentre Study
Brief Title: Predicting Morbidity and Mortality in Elderly Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital of Navarra (Other)
Collaborators: Hospital Universitario Alava (Unknown); Hospital de Cruces (Other); Hospital de Basurto (Other); Hospital Donostia (Other); Hospital San Pedro de Logroño (Other)
Responsible Party: Principal Investigator, Ines Eguaras, Principal Investigator, Hospital of Navarra
Other Study IDs: Hospital Universitario Navarra
Record Dates: First submitted 2021-12-27; First posted 2022-01-31 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Surgery--Complications
Keywords: Elderly; urgent abdominal surgery; 30-day mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Hospital Universitario de Álava, Spain: large hospitals (>200 beds) with wards admitting older surgical patients where (a) electronic medical records are available, (b) have staff committed to recruiting a minimum of 100 participants with complete follow-up, and (c) give consent for the Lead statistician in Spain to access de-identified data for aggregated analysis.
- Hospital Universitario de Basurto, Spain: large hospitals (>200 beds) with wards admitting older surgical patients where (a) electronic medical records are available, (b) have staff committed to recruiting a minimum of 100 participants with complete follow-up, and (c) give consent for the Lead statistician in Spain to access de-identified data for aggregated analysis.
- Hospital Universitario de Cruces, Spain: large hospitals (>200 beds) with wards admitting older surgical patients where (a) electronic medical records are available, (b) have staff committed to recruiting a minimum of 100 participants with complete follow-up, and (c) give consent for the Lead statistician in Spain to access de-identified data for aggregated analysis.
- Hospital Universitario de Donostia, Spain: large hospitals (>200 beds) with wards admitting older surgical patients where (a) electronic medical records are available, (b) have staff committed to recruiting a minimum of 100 participants with complete follow-up, and (c) give consent for the Lead statistician in Spain to access de-identified data for aggregated analysis.
- Hospital San Pedro (Logroño), Spain: large hospitals (>200 beds) with wards admitting older surgical patients where (a) electronic medical records are available, (b) have staff committed to recruiting a minimum of 100 participants with complete follow-up, and (c) give consent for the Lead statistician in Spain to access de-identified data for aggregated analysis.
- Hospital of Navarra, Spain: large hospitals (>200 beds) with wards admitting older surgical patients where (a) electronic medical records are available, (b) have staff committed to recruiting a minimum of 100 participants with complete follow-up, and (c) give consent for the Lead statistician in Spain to access de-identified data for aggregated analysis.

SUMMARY:
This proposed multicentre study builds on the findings of our recent validation of USEM and mCriSTAl predictive tools in a single centre at the Complejo Hospitalario de Navarra, whose results were recently published (https://europepmc.org/article/med/33111261). By expanding to a multicentre cohort and comparing to a third instrument, the investigators aim to examine the independent validity and generalizability of three scores and investigate potential for simplification of the prediction with anticipated greater accuracy. The ultimate goal is to determine whether these predictive tool can be used to assist surgical decision-making about older patients with expected poorer prognosis or high risk of death in the short term.

DETAILED DESCRIPTION:
Eligible institutions: large hospitals (>200 beds) with wards admitting older surgical patients where (a) electronic medical records are available, (b) have staff committed to recruiting a minimum of 100 participants with complete follow-up, and (c) give consent for the Lead statistician in Spain to access de-identified data for aggregated analysis.

Procedures: Recruitment is anticipated to take 6-12 months and will be conducted prospectively after screening by non-specialist hospital staff (junior doctors, medical students, nurses) confirms eligibility. The 3-month follow-up for outcomes will include completion of a standard questionnaire/form via either review of clinical record, access to death records (where applicable), or telephone call to families/proxy/next of kin/person responsible at 3 months after initial recruitment.

Findings will be published in aggregated and anonymized form, but if the sample from individual participating institutions is large enough, hospital-specific profiles can be delivered in identifiable form to relevant hospitals for the benefit of clinicians and service administrators.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥65 years.
* Present in the ED with acute abdominal pathology that requires urgent abdominal surgery

Exclusion Criteria:

* Patients who receive non-operative management
* Informed consent form not signed by patient or their proxy

Ages: 65 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: large hospitals (>200 beds) with wards admitting older surgical patients where (a) electronic medical records are available, (b) have staff committed to recruiting a minimum of 100 participants with complete follow-up, and (c) give consent for the Lead statistician in Spain to access de-identified data for aggregated analysis.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of postoperative mortality | 30 day
  prediction of the individual tools as ascertained from the official mortality records
Number of postoperative mortality | 90 day
  prediction of the individual tools as ascertained from the official mortality records
In-hospital surgery-related adverse events | 30 day
  Defined by the Clavien-Dindo classification

SECONDARY OUTCOMES:
validity of the score | 30-day
  Discrimination and calibration of the new tool, compared to the: m CRISTAL, USEM, NELA
validity of the score | 90-day
  Discrimination and calibration of the new tool, compared to the: m CRISTAL, USEM, NELA

CONTACTS AND LOCATIONS:
Locations (1):
- UPNA, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No